CLINICAL TRIAL: NCT02603913
Title: Oxidative Stress and Endothelial Function in Pregnancy Complications: Development of a New Screening Algorithm
Brief Title: Oxidative Stress and Endothelial Function in Pregnancy Complications
Acronym: ENDOPREG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Ziekenhuis Oost-Limburg (Other); Maastricht University Medical Center (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof Yves Jacquemyn, Professor, Universiteit Antwerpen
Other Study IDs: UZA-Endopreg-2015-1
Record Dates: First submitted 2015-10-18; First posted 2015-11-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy Complications; Endothelial Dysfunction
Keywords: Pre-eclampsia; Pregnancy induced hypertension; Preterm birth; Intra-uterine growth restriction; Oxidative stress
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and placenta samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal pregnancy: Normal uncomplicated pregnancy
- Pre-eclampsia: Hypertension (>140 mmHg systolic or >90 mmHg diastolic) developing after 20 weeks gestation and the coexistence of one or more of the following new onset conditions:
  1. Proteinuria (>300 mg/day)
  2. Other maternal organ dysfunction
     * renal insufficiency (creatinine >90 μmol/L)
     * liver involvement (elevated transaminases - and/or severe right upper quadrant or epigastric pain)
     * neurological complications (eclampsia, altered mental status, blindness, stroke, hyperreflexia when accompanied by clonus, severe headaches when accompanied by hyperreflexia, persistent visual scotomata)
     * hematological complications (thrombocytopenia, disseminated intravascular coagulation, hemolysis)
  3. Uteroplacental dysfunction
- Pregnancy induced hypertension: New onset of hypertension (>140 mmHg systolic or >90 mmHg diastolic) after 20 weeks gestation, without proteinuria, in a previously normotensive woman.
- Preterm birth: Babies born alive before 37 weeks of pregnancy are completed.
- Intra-uterine growth restriction: Moderate IUGR is an estimated fetal weight and / or abdominal circumference < 10th percentile for its gestational age Severe IUGR is an EFW (estimated fetal weight) and/ or AC (abdominal circumference) < 5th percentile for its gestational age

SUMMARY:
Pregnancy complications like pre-eclampsia (PE), pregnancy induced hypertension (PIH), intra-uterine growth restriction (IUGR) and preterm labor (PTL), (i.e. the major part of complications in pregnancy) are related to an impaired endothelial function. Endothelial dysfunction accounts for altered vascular reactivity, activation of the coagulation cascade and loss of vascular integrity. Nitric oxide (NO), a free radical molecule derived from L-Arginine by NOS (Nitric Oxide Synthase), is an endogenous endothelium-derived relaxing factor influencing endothelial function. In the placental circulation, endothelial release of NO dilates the fetal placental vascular bed and thus ensures feto-maternal exchange. The impaired endothelial function in pregnancy complications originates from production of inflammatory and cytotoxic factors by the ischemic placenta and results in oxidative stress and an altered bioavailability of NO. Measurement of endothelial function using peripheral artery tonometry and determination of ROS (reactive oxygen species) and RNS (reactive nitrogen species) using Electron Paramagnetic Resonance (EPR) gives an idea of the oxidative stress that took place and the degree of endothelial dysfunction that occurred during pregnancy.

DETAILED DESCRIPTION:
INTRODUCTION. In normal pregnancy vascular remodelling of the maternal uterine spiral arteries occurs. Trophoblast cells invade the spiral arterioles within the first 12 weeks of pregnancy and replace the muscular wall of the vessels converting them into wide bore, low resistance, large capacity vessels, a process normally completed by 20 weeks gestation. The pathogenesis of generalized endothelial dysfunction in complicated pregnancies is subdivided into two phases. The first phase exists of a poor trophoblast invasion of the spiral arteries during the placentation process, causing failure to transform the placental bed arteries from high to low resistance vessels. This results in local ischemia, reperfusion damage and oxidative stress. The local damage activates the second phase where enhanced production of anti-angiogenic factors and oxidative stress products results in systemic inflammation, endothelial activation and decreased endothelial nitric oxide. In case the endothelial damage is most outspoken, thrombotic micro-angiopathy is induced with platelet-fibrin thrombi in micro-vessels. The angiopathy results in consumption of circulating platelets, causes hemolysis in affected micro-vessels and reduces portal blood flow in the liver, finally resulting in periportal necrosis, a condition seen in severe pre-eclampsia (PE).

HYPOTHESIS.

* Increased oxidative stress and endothelial dysfunction are present early in pregnancy when pregnancy complications will develop later on.
* Oxidative stress and endothelial dysfunction are not entirely independent from each other and can be measured.
* Oxidative stress can be reduced and endothelial function can be improved by interventions that will reduce the risk of developing pregnancy complications.

Thus: measurement and integration in an algorithm of oxidative stress and endothelial function in early pregnancy will allow us to determine which pregnancies will benefit from preventive interventions. This selection will optimize targeted interventions on high risk pregnancies without overtreatment of others.

METHODOLOGY

1. Study design 1.1. Single center prospective longitudinal study For the first part of the study, the investigators propose a prospective longitudinal design. Pregnant women in their first trimester of pregnancy, will be eligible and will be followed throughout pregnancy and until 6 months postpartum.

   1.2. Multicenter matched case-control study The second part is a case control study where patients with pregnancies complicated by PIH / PE / preterm birth / IUGR will be compared to normotensive controls, matched for maternal and gestational age, parity, smoking behavior, BMI and ethnic group. Patients will be followed throughout (the rest of their) pregnancy and until 6 months postpartum. The patients in this study will be included in UZA, Erasmus MC, Maastricht UMC, ZOL (Ziekenhuis Oost-Limburg).
2. Description of investigations 2.1 Endothelial function (RHI): The reactive hyperemia index is measured using peripheral artery tonometry (PAT) (endoPAT®, Itamar). The tonometer consists of a finger- mounted probe plethysmograph, capable of sensing volume changes in the vessels of the index fingers. It is a non-operator-dependent and thus reproducible technique. Sensors are placed at the fingertips of the index fingers.

Suprasystolic occlusion of the non-dominant upper arm, at 200mmHg or 60 mmHg above systolic blood pressure, will be obtained using a cuff. After upper-arm occlusion the response to reactive hyperemia will be measured. The contralateral (dominant) arm is used as control, to correct for systemic effects.

2.2 Arterial stiffness (PWV, PWA): Pulse wave velocity and pulse wave analysis will be calculated using the Sphygmocor system ® (Atcor Medical, West Ryde, Australia). To calculate PWV, two pressure waveforms must be measured at a known distance apart and the distance between measurement sites is divided by the propagation time. Aortic PWV is measured by carotid-femoral PWV (cfPWV) as it is the 'gold standard' measurement of the stiffness of the aorta. Measurements of cfPWV will be performed using a pressure tonometer to transcutaneously record the pressure pulse waveform in the underlying artery. The tonometer contains a micromanometer that provides a very accurate recording of the pressure within the artery. The carotid and femoral PWV will be assessed by gently compressing respectively the carotid artery and the femoral artery with the tip of the tonometer at the site of maximal pulsation. The Sphygmocor device will automatically calculate the cfPWV. PWA will calculate AIx by placing the tonometer at the radial artery (site of maximum pulsation). A generalized transfer function will derive the aortic pressure waveform from the radial artery waveform. From the aortic pressure waveform, the augmentation pressure (AP) and augmentation index (AIx) can be calculated. The AP (ΔP) is defined as the height of the late systolic peak above the inflection point on the waveform. The AIx is defined as AP expressed as a percentage of the aortic PP. As AIx is affected by heartrate, it will be standardized to a heart rate of 75 bmp (AIx-75).

2.3 Pulsatility index uterine artery (PI UA) and fetal biometry: Uterine artery Doppler examinations will be performed using trans-abdominal color directed pulsed wave Doppler (Voluson, GE Healthcare Technologies, USA). PI of both uterine arteries will be obtained on either side of the cervix before 14 weeks' gestation and at the apparent crossover with the external iliac arteries after 14 weeks. At the same moment basic fetal biometry parameters will be measured: bi-parietal diameter, head circumference, abdominal circumference, femur length and expected fetal weight using Hadlocks formula.

2.4 NLR and MPV: Performing a complete blood count, NLR, MPV and platelet count will be obtained using a ADVIA 120 Hematology System (Siemens healthcare, Germany).

2.5 Automated blood pressure measurement: SBP (systolic blood pressure), DBP (diastolic blood pressure) and MAP (mean arterial pressure) after 10 minutes rest in a sitting position, will be measured using a Mindray VS 900 monitor (Mindray, China).

2.6 Oxidative stress 2.6.1 Electron paramagnetic resonance: NO and O2∙- EPR (electron paramagnetic resonance) is derived from magnetic resonance spectroscopy and uses microwave radiation to detect molecules with an unpaired electron number, like radicals. When an magnetic field is created by the EPR spectrometer, all radicals will align. The EPR spectrometer sends out a radio frequent microwave, causing the electrons to jump from a low to a high energy state. This energy absorption can be measured and is directly correlated to the amount of free radicals in the sample. A 'spin trap' will be added to scavenge the very reactive radicals and to prolong their half live. The concentration of NO will be determined using an Iron-DETC (Fe(II)DETC2 (iron(II)diethyldithiocarbamaat) solution. The spin probe for the determination of O2∙- (superoxide) in maternal serum is CMH (1-Hydroxy-3-methoxycarbonyl-2,2,5,5-tetramethylpyrrolidine) and in placental tissue this is ascorbic acid (Vitamin C). Vitamin C has an anti-oxidative effect and is abundantly present in the human body. O2∙- reacts easily with vitamin C to form the ascorbic radical. This ascorbic radical is a measure for the O2∙- concentration in placental tissue. Placental tissue will be investigated at the time of delivery, maternal serum at week 9, week 28, at delivery and 6 months post-partum.

2.6.2 Western blot analyse: ONOO-, eNOS en iNOS NO and O2∙- react to form ONOO-. The ONOO- production will be indirectly measured in placental tissue via tyrosine nitration. Nitrotyrosine arises when ONOO- reacts with tyrosine in proteins and can be quantified in placental tissue with Western blotting using anti-nitrotyrosine antibodies. NO is formed out of L-Arginine by NOS (Nitric Oxide Synthase). This reaction is regulated by VEGF (Vascular endothelial growth factor), an endothelial mitogen that has an important function in the proliferation of endothelial cells and in angiogenesis. VEGF stimulates eNOS (endothelial NOS) and induces therefore NO production. Placental ischemia will increase VEGF-production and thus raise NO-production, as an compensatory mechanism to guarantee sufficient feto-maternal transfusion. In an oxidative environment, the lack of NOS-stabilizing factors results in NOS-uncoupling. NOS-coupling causes a shift from NO production to O2∙- production. This maintains an oxidative setting. iNOS (inducible NOS) production is induced by cytokines and endotoxins during inflammatory conditions. Monoclonal antibodies will determine concentrations of eNOS and iNOS in placental tissue.

STATISTICAL ANALYSIS

1. Sample size calculation 1.1. Single center prospective longitudinal study For the physiologic study of the RHI in pregnancy the investigators calculated that for a 95% confidence interval, a population standard deviation of 0.5 (as described in other populations for RHI) and a tolerable standard error of the mean (SEM) value of 0.1, 97 women have to be followed. Taking at least a 10% dropout into account the starting sample size will be 110 women.

   1.2. Multicenter matched case-control study In a pilot study by Yinon [Yinon, 2006] the reactive hyperemia index (RHI) in normotensive pregnancies was 1.8, and in PE 1.5; in most populations standard deviation is 0.5. For 80% power and a two sided α = 0.05 and considering a 0.3 difference clinically relevant, the sample size for each group would be 44; which will be considered the sample size for the cross-sectional study comparing PE (44), PIH (44), IUGR (44) and preterm birth (44) with normotensive controls (44).
2. Descriptive statistics and data analysis 2.1. Single center prospective longitudinal study For the physiologic study of the RHI in pregnancy the investigators will calculate the reference values and 95% confidence interval. Longitudinal data will be plotted and a linear mixed-effects model with random intercept will be fitted. Percentiles for RHI and PWV will be calculated based on this model. Correlation coefficients between baseline RHI, PWV, UA Doppler PI, fetal biometry, NLR, MPV, MAP, birth-weight percentile and EDCs will be analyzed.

2.2. Multicenter matched case-control study RHI, PWV, UA Doppler PI, fetal biometry, NLR, MPV, MAP, birth-weight and EDCs and other continuous variables in hypertensive versus non hypertensive pregnancies will be tested for normality using the Shapiro Wilk Test. If there is normality, they will be expressed as mean, standard deviations and 95% confidence intervals and compared using two sided T test. If not, they will be expressed as median and interquartile ranges and compared using Mann Whitney U Test.

ELIGIBILITY:
Inclusion Criteria:

* Prospective longitudinal study:

  * Pregnant women ≥ 18 years old with a singleton pregnancy
* Case-control study:

  * Pregnant women ≥ 18 years old with a singleton pregnancy and > 20 weeks of pregnancy.
  * Cases: Pre-eclampsia, PIH, IUGR, Preterm birth (cfr groups)

Exclusion criteria:

* gestational diabetes
* multiple pregnancies
* fetal abnormalities
* hypercholesterolemia
* renal disease
* auto-immune disorders
* connective tissue disease
* intake of low-dose aspirin or vitamin C supplements (>500mg/day)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be included at one of the participating tertiary obstetrical centers (UZA, ZOL, Erasmus MC, MUMC).
  They will be included at the beginning of pregnancy in the longitudinal studies. In the case-control study, they will be included at the moment of diagnosis and compared to normotensive controls, matched for maternal and gestational age, parity, smoking behavior, BMI and ethnic group.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress. Measurement of nitric oxide and eNOS in placental tissue and superoxide in maternal serum using EPR and western blotting. | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study: To evaluate the oxidative stress profile in normal pregnancies.
  Multicenter matched case-control study: To compare the oxidative stress profile in normal versus complicated pregnancies.

SECONDARY OUTCOMES:
Endothelial function (using Endopat®) | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study: To evaluate endothelial function in normal pregnancies.
  Multicenter matched case-control study: To compare endothelial function in normal versus complicated pregnancies.
  To relate endothelial function (using Endopat ®) to nitric oxide/eNOS/superoxide concentration (using EPR and Western Blotting).
Arterial stiffness (Pulse wave velocity, pulse wave analysis using Sphygmocor ®). | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study: To evaluate arterial stiffness in normal pregnancies.
  Multicenter matched case-control study: To compare arterial stiffness in normal versus complicated pregnancies.
  To relate Arterial stiffness (using Sphygmocor ®) to nitric oxide/eNOS/superoxide concentration (using EPR and Western Blotting).
Pregnancy outcome | Pregnancy - 6 months postpartum
  Pregnancy outcome will be determined using the diagnostic criteria described in 'groups and interventions'.
  Single center prospective longitudinal study and multicenter matched case-control study.
  To relate oxidative stress profile to pregnancy outcome.
Pulsatility index uterine artery (using doppler ultrasound). | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study and multicenter matched case-control study.
Mean platelet volume (MPV (fL)) | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study and multicenter matched case-control study.
Neutrophil-lymphocyte ratio (NLR) | Pregnancy - 6 months postpartum
  Single center prospective longitudinal study and multicenter matched case-control study.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique AM Mannaerts, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Chen X, Scholl TO. Maternal biomarkers of endothelial dysfunction and preterm delivery. PLoS One. 2014 Jan 22;9(1):e85716. doi: 10.1371/journal.pone.0085716. eCollection 2014. PMID 24465662
- [Background] Yinon D, Lowenstein L, Suraya S, Beloosesky R, Zmora O, Malhotra A, Pillar G. Pre-eclampsia is associated with sleep-disordered breathing and endothelial dysfunction. Eur Respir J. 2006 Feb;27(2):328-33. doi: 10.1183/09031936.06.00010905. PMID 16452588
- [Background] Bhavina K, Radhika J, Pandian SS. VEGF and eNOS expression in umbilical cord from pregnancy complicated by hypertensive disorder with different severity. Biomed Res Int. 2014;2014:982159. doi: 10.1155/2014/982159. Epub 2014 May 14. PMID 24959596
- [Background] Sikkema JM, van Rijn BB, Franx A, Bruinse HW, de Roos R, Stroes ES, van Faassen EE. Placental superoxide is increased in pre-eclampsia. Placenta. 2001 Apr;22(4):304-8. doi: 10.1053/plac.2001.0629. PMID 11286565
- [Background] Tranquilli AL, Dekker G, Magee L, Roberts J, Sibai BM, Steyn W, Zeeman GG, Brown MA. The classification, diagnosis and management of the hypertensive disorders of pregnancy: A revised statement from the ISSHP. Pregnancy Hypertens. 2014 Apr;4(2):97-104. doi: 10.1016/j.preghy.2014.02.001. Epub 2014 Feb 15. No abstract available. PMID 26104417
- [Derived] Mannaerts D, Faes E, Gielis J, Van Craenenbroeck E, Cos P, Spaanderman M, Gyselaers W, Cornette J, Jacquemyn Y. Oxidative stress and endothelial function in normal pregnancy versus pre-eclampsia, a combined longitudinal and case control study. BMC Pregnancy Childbirth. 2018 Feb 27;18(1):60. doi: 10.1186/s12884-018-1685-5. PMID 29482567